CLINICAL TRIAL: NCT01474434
Title: A Randomized, Double-blind, Placebo Controlled Study to Assess the Efficacy of LCQ908 on Cardiovascular Risk
Brief Title: Efficacy of LCQ908 on Cardiovascular Risk
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated based on interim analysis. See detailed description.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CLCQ908A2213
Record Dates: First submitted 2011-11-09; First posted 2011-11-18 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Artery Disease; Hypertriglyceridemia
Keywords: coronary artery disease,; LCQ908,; hyperlipidemia,; hypertriglyceridemia,; pradigastat
MeSH Terms: conditions — Coronary Artery Disease; Hypertriglyceridemia; Hyperlipidemias | interventions — pradigastat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Pradigastat (LCQ908) followed by placebo (Experimental): Pradigastat 80 mg (4 x 20-mg tablets) loading dose daily for three days followed by pradigastat 20 mg (2 x 10-mg tablets) daily for two days followed by a 30-day washout period in between followed by 5-day placebo treatment
  Interventions: Drug: pradigastat (LCQ908); Drug: Placebo
- Placebo followed by pradigastat (LCQ908) (Experimental): Placebo (5-day treatment period) followed by a 30-day washout period followed by pradigastat 80 mg (4 x 20-mg tablets) loading dose daily for three days followed by p20 mg (2 x 10-mg tablets) daily for two days
  Interventions: Drug: pradigastat (LCQ908); Drug: Placebo

INTERVENTIONS:
Drug: pradigastat (LCQ908) — pradigastat tablets were supplied to the investigators at dose strengths of 10 mg and 20 mg as individual patient packs.
  Other Names: Pradigastat
Drug: Placebo — matching placebo tablets

SUMMARY:
This is a study designed to evaluate the potential for the pradigastat (LCQ908) to impact cardiovascular risk.

DETAILED DESCRIPTION:
This study had 2 parts. Part A was a multicenter, double-blind, randomized, placebo-controlled, non-confirmatory crossover study assessing response to a high-fat meal challenge in the setting of pradigastat versus placebo. Part A had 2 cohorts i.e. Cohort 1 patients with stable coronary artery disease and hypertriglyceridemia and Cohort 2 patients with asymptomatic non-obstructive coronary artery disease or elevated coronary heart disease risk and hypertriglyceridemia.

Part B was a double blinded phase designed to assess response to three months of chronic treatment with pradigastat versus placebo on a normal diet.

The trial was terminated after the interim analysis of Part A, Cohort 1. The interim analysis results indicated that the high-fat meal challenge did not induce any impairment on either myocardial perfusion reserve index (MPRi) or exercise treadmill performance. Part B was never started.

ELIGIBILITY:
Inclusion Criteria:

* History of coronary artery disease
* Elevated triglycerides
* On medication to help lower cholesterol

Exclusion Criteria:

* Poorly controlled diabetic patients and/or change in diabetic medication within 12 weeks of screening
* History of myocardial infarction (heart attack) within 6 months of screening
* History of a procedure to open a blocked coronary artery within 12 months of enrollment
* History of Coronary Artery Bypass Graft (CABG) surgery
* History of congestive heart failure
* History of significant heart valve disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Pasadena, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was terminated upon Part A interim analysis. Total 41 patients randomized to Part A i.e.17 patients in cohort 1 and 24 patients in Cohort 2.
Groups:
- Part A, Cohort 1: Pradigastat (LCQ908) Followed by Placebo: Cohort 1 consisted of patients with evidence of stable symptomatic or obstructive coronary artery disease and mild to moderate hypertriglyceridemia. All patients who randomized to this sequence received pradigastat 80 mg (4 x 20-mg tablets) loading dose daily for three days followed by pradigastat 20 mg (2 x 10-mg tablets) daily for two days followed by a 30-day washout period in between followed by 5-day placebo treatment
- Part A, Cohort 1: Placebo Followed by Pradigastat (LCQ908): Cohort 1 consisted of patients with evidence of stable symptomatic or obstructive coronary artery disease and mild to moderate hypertriglyceridemia. All patients who randomized to this sequence received Placebo (5-day treatment period) followed by a 30-day washout period followed by pradigastat 80 mg (4 x 20-mg tablets) loading dose daily for three days followed by 20 mg (2 x 10-mg tablets) daily for two days
- Part A, Cohort 2: Pradigastat (LCQ908) Followed by Placebo: Cohort 2 consisted of patients with stable asymptomatic non-obstructive coronary artery disease or coronary heart disease risk equivalents and mild to moderate hypertriglyceridemia.. All patients who randomized to this sequence received pradigastat 80 mg (4 x 20-mg tablets) loading dose daily for three days followed by pradigastat 20 mg (2 x 10-mg tablets) daily for two days followed by a 30-day washout period in between followed by 5-day placebo treatment
- Part A, Cohort 2: Placebo Followed by Pradigastat (LCQ908): Cohort 2 consisted of patients with stable asymptomatic non-obstructive coronary artery disease or coronary heart disease risk equivalents and mild to moderate hypertriglyceridemia. All patients who randomized to this sequence received Placebo (5-day treatment period) followed by a 30-day washout period followed by pradigastat 80 mg (4 x 20-mg tablets) loading dose daily for three days followed by 20 mg (2 x 10-mg tablets) daily for two days
Period: Treatment Period 1 (5 Days [Day 1 - 5])
Arm/Group | Part A, Cohort 1: Pradigastat (LCQ908) Followed by Placebo | Part A, Cohort 1: Placebo Followed by Pradigastat (LCQ908) | Part A, Cohort 2: Pradigastat (LCQ908) Followed by Placebo | Part A, Cohort 2: Placebo Followed by Pradigastat (LCQ908)
Started | 8 | 9 | 11 | 13
Completed | 7 | 9 | 10 | 11
Not Completed | 1 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Protocol deviation | 1 | 0 | 0 | 0
Period: Treatment Period 2(5 Days[Day 36 - 40])
Arm/Group | Part A, Cohort 1: Pradigastat (LCQ908) Followed by Placebo | Part A, Cohort 1: Placebo Followed by Pradigastat (LCQ908) | Part A, Cohort 2: Pradigastat (LCQ908) Followed by Placebo | Part A, Cohort 2: Placebo Followed by Pradigastat (LCQ908)
Started | 7 | 9 | 10 | 11
Completed | 7 | 9 | 10 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all patients who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Cohort 1: Pradigastat (LCQ908) Followed by Placebo | Part A, Cohort 1: Placebo Followed by Pradigastat (LCQ908) | Part A, Cohort 2: Pradigastat (LCQ908) Followed by Placebo | Part A, Cohort 2: Placebo Followed by Pradigastat (LCQ908) | Total
Number analyzed (Participants) | 8 | 9 | 11 | 13 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (6.67) | 58.4 (8.79) | 56.7 (9.79) | 56.1 (8.85) | 57.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 6 | 16
  Male | 6 | 5 | 7 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Myocardial Perfusion Reserve Index (MPRi) Overall Mean (Part A, Cohort 1)
Description: MPRi (myocardial perfusion reserve index) is a measure of coronary microvascular function. Myocardial perfusion scans using 0.05 mmol/kg of gadolinium contrast were acquired at rest and under stress (pharmacological stress induced with adenosine 140 μg/kg/min for three minutes). An independent central reader performed the cardiac image analysis of all time points including the calculation of the myocardial perfusion reserve index from the ratio of the global stress myocardial blood flow divided by the resting blood flow values. Higher/increased index indicates improved flow/better outcome. This primary endpoint was only for Part A, Cohort 1 patients.
Time Frame: Baseline, and on day 5 of each of the two treatment periods
Population: Efficacy analysis set - Patients who took > 80% of study drug as assessed by drug accountability, had no major protocol deviations, and had a valid assessment of MPRi at both baseline and post-treatment visits. Patients who had no baseline or post-treatment MPRi data in 1 of 2 periods were excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: myocardial perfusion reserve index
Groups:
- Part A, Cohort 1: Pradigastat (LCQ908): Cohort 1 consisted of patients with evidence of stable symptomatic or obstructive coronary artery disease and mild to moderate hypertriglyceridemia. All randomized patients who received pradigastat in either of 2 treatment period.
- Part A, Cohort 1: Placebo: Cohort 1 consisted of patients with evidence of stable symptomatic or obstructive coronary artery disease and mild to moderate hypertriglyceridemia. All randomized patients who received matching placebo in either of 2 treatment period
Arm/Group | Part A, Cohort 1: Pradigastat (LCQ908) | Part A, Cohort 1: Placebo
Number analyzed (Participants) | 13 | 12
myocardial perfusion reserve index | -0.22 (0.24) | 0.32 (0.24)

2. Primary Outcome: Change From Baseline in Total Exercise Duration (Part A, Cohort 1)
Description: Total exercise duration was the elapsed time between the start of exercise and termination of exercise for severe angina, dyspnea or extreme fatigue. This primary endpoint was only for Part A, Cohort 1 patients.
Time Frame: Baseline and on day 5 of each of the two treatment periods
Population: Efficacy analysis set- Patients who took > 80% of study drug as assessed by drug accountability, had no major protocol deviations, and had a valid assessment of total exercise duration at both baseline and post-treatment visits. Patients who had no baseline or post-treatment exercise duration data in 1 of 2 periods were excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: minute
Arm/Group | Part A, Cohort 1: Pradigastat (LCQ908) | Part A, Cohort 1: Placebo
Number analyzed (Participants) | 11 | 14
minute | -1.52 (0.46) | -1.00 (0.40)

3. Primary Outcome: Time to Onset of Angina (Part A, Cohort 1)
Description: Time to onset of angina was defined as the elapsed time between the start of exercise and the onset of anginal chest pain as reported by the patient and recorded by the performing investigator.
Time Frame: Baseline and on day 5 of each of the two treatment periods
Population: The study was terminated based on the interim analysis after patients completed Part A. This outcome measure was not part of interim analysis; hence it is not done. .
Arm/Group | Part A, Cohort 1: Pradigastat (LCQ908) | Part A, Cohort 1: Placebo
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Time to Onset of Exercise-induced Ischemia(Part A, Cohort 1)
Description: Exercise-induced ischemia was defined as the new development of horizontal or down-sloping ST-segment depression (≥ 1mm at 60 milliseconds after the J point) versus baseline tracings.
Time Frame: Baseline and on day 5 of each of the two treatment periods
Population: as for outcome 3
Arm/Group | Part A, Cohort 1: Pradigastat (LCQ908) | Part A, Cohort 1: Placebo
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Aortic Plaque Inflammation (Part B)
Description: This endpoint was palnned for analysis on Part B patients which was never started becasue study got terminated on Part A interim analysis.
Time Frame: Baseline and on treatment day 85 +/- 3 days
Population: The study was terminated based on the interim analysis after patients completed Part A. Part B of the study was never started.
Arm/Group | Part B: Pradigastat (LCQ908) | Part B: Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Adverse Events (Part A, Cohort 1)
Time Frame: approximately 40 days
Population: The safety analysis set included all patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Part A, Cohort 1: Pradigastat (LCQ908) | Part A, Cohort 1: Placebo
Number analyzed (Participants) | 17 | 17
Participants
  Any Adverse Events | 16 | 6
  Serious Adverse Events | 0 | 0
  Death | 0 | 0

7. Secondary Outcome: Number of Participants With Adverse Events (Part A, Cohort 2)
Time Frame: approximately 40 days
Population: The safety analysis set included all patients who received at least one dose of study drug.
Measure: Number; unit: Participants
Groups:
- Part A, Cohort 2: Pradigastat (LCQ908): Cohort 2 consisted of patients with stable asymptomatic non-obstructive coronary artery disease or coronary heart disease risk equivalents and mild to moderate hypertriglyceridemia.. All randomized patients who recieved pradigastat in either of 2 treatment period.
- Part A, Cohort 2: Placebo: Cohort 2 consisted of patients with stable asymptomatic non-obstructive coronary artery disease or coronary heart disease risk equivalents and mild to moderate hypertriglyceridemia. All randomized patients who received matching placebo in either of 2 treatment period
Arm/Group | Part A, Cohort 2: Pradigastat (LCQ908) | Part A, Cohort 2: Placebo
Number analyzed (Participants) | 24 | 24
Participants
  Any Adverse Events | 22 | 15
  Serious Adverse Events | 0 | 1
  Death | 0 | 0

8. Secondary Outcome: Postprandial Triglycerides (Part A, Cohort 1)
Description: For both each treatment period, postprandial triglycerides were measured on Day 5 i.e. on 0 hour(before breakfast), two hours and four hours post high-fat breakfast. Results are from an ANCOVA model on change from baseline in the log domain with log(baseline), treatment, sequence and period as fixed effects. Baseline is the Day -1 value within period. The data reported is ratio of geometric mean between post-treatment and baseline data.
Time Frame: 0 hour (before breakfast), 2 and 4 hours post high-fat breakfast on day 5
Population: The efficacy analysis set included all patients who took more than 80% of study medication as assessed by drug accountability, had no major protocol deviations, and had a valid assessment of the primary efficacy variables at both baseline and post treatment visits.
Measure: Geometric Mean (Standard Error); unit: ratio
Arm/Group | Part A, Cohort 1: Pradigastat (LCQ908) | Part A, Cohort 1: Placebo
Number analyzed (Participants) | 16 | 16
ratio
  Day 5 Hr 0 | 1.15 (1.08) | 0.97 (1.08)
  Day 5 Hr 2 | 1.21 (1.08) | 1.40 (1.07)
  Day 5 Hr 4 | 1.29 (1.09) | 1.71 (1.08)

9. Secondary Outcome: Postprandial Triglycerides (Part A, Cohort 2)
Description: For both each treatment period, postprandial triglycerides were measured on Day 5 i.e. on 0 hour (before breakfast), two hours and four hours post high-fat breakfast. Results are from an ANCOVA model on change from baseline in the log domain with log(baseline), treatment, sequence and period as fixed effects. Baseline is the Day -1 value within period. The data reported is ratio of geometric mean between post-treatment and baseline data.
Time Frame: 0 hour (before breakfast), 2 and 4 hours post high-fat breakfast on day 5
Population: as for outcome 8
Measure: Geometric Mean (Standard Error); unit: ratio
Arm/Group | Part A, Cohort 2: Pradigastat (LCQ908) | Part A, Cohort 2: Placebo
Number analyzed (Participants) | 19 | 19
ratio
  Day 5 Hr 0 | 1.16 (1.08) | 1.09 (1.08)
  Day 5 Hr 2 | 1.15 (1.07) | 1.38 (1.07)
  Day 5 Hr 4 | 1.14 (1.08) | 1.56 (1.08)

10. Secondary Outcome: Pharmacokinetics of Pradigastat (LCQ908): Plasma Concentration (Part A)
Time Frame: Part A: Day 4 and day 5 of each treatment period
Population: The study was terminated based on the interim analysis on Part A, Cohort 1 after patients completed Part A. The analysis of this assessment was not part of interim analysis; hence it is not done.
Arm/Group | Part A, Cohort 1: Pradigastat (LCQ908) | Part A, Cohort 1: Placebo | Part A, Cohort 2: Pradigastat (LCQ908) | Part A, Cohort 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Other Related Lipid Parameters (Part A)
Time Frame: Baseline, day 4 and day 5 of each treatment period
Population: as for outcome 10
Arm/Group | Part A, Cohort 1: Pradigastat (LCQ908) | Part A, Cohort 1: Placebo | Part A, Cohort 2: Pradigastat (LCQ908) | Part A, Cohort 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Interleukin-6 (IL-6) Level (Part A)
Time Frame: Baseline, day 4 and day 5, of each treatment period
Population: as for outcome 10
Arm/Group | Part A, Cohort 1: Pradigastat (LCQ908) | Part A, Cohort 1: Placebo | Part A, Cohort 2: Pradigastat (LCQ908) | Part A, Cohort 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: C-reactive Protein (CRP) Level (Part A)
Time Frame: Baseline, day 4 and day 5, of each treatment period
Population: as for outcome 10
Arm/Group | Part A, Cohort 1: Pradigastat (LCQ908) | Part A, Cohort 1: Placebo | Part A, Cohort 2: Pradigastat (LCQ908) | Part A, Cohort 2: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Adiponectin Level ( Part B)
Time Frame: Part B; Baseline, day 15, day 43 and day 85
Population: The study was terminated based on the interim analysis on Part A, cohort 1 after patients completed Part A. Part B of the study was not commenced.
Arm/Group | Part B: Pradigastat (LCQ908) | Part B: Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The safety analysis set included all patients who received at least one dose of study drug.
Arm/Group | Part A, Cohort 1: Pradigastat (LCQ908) | Part A, Cohort 1: Placebo | Part A, Cohort 2: Pradigastat (LCQ908) | Part A, Cohort 2: Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/24 | 1/24
Other Adverse Events (participants affected / at risk) | 16/17 | 6/17 | 22/24 | 13/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Cohort 1: Pradigastat (LCQ908) (N=17) | Part A, Cohort 1: Placebo (N=17) | Part A, Cohort 2: Pradigastat (LCQ908) (N=24) | Part A, Cohort 2: Placebo (N=24)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Cohort 1: Pradigastat (LCQ908) (N=17) | Part A, Cohort 1: Placebo (N=17) | Part A, Cohort 2: Pradigastat (LCQ908) (N=24) | Part A, Cohort 2: Placebo (N=24)
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 5 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 15 | 1 | 21 | 8
Nausea (Gastrointestinal disorders) | 9 | 1 | 13 | 5
Vomiting (Gastrointestinal disorders) | 6 | 0 | 6 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 2 | 0 | 4 | 1
Polyuria (Renal and urinary disorders) | 1 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated based on the interim analysis on Part A, Cohort 1 after patients completed Part A. Part B was not conducted. Not all the planned assessments were completed due to the termination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.